CLINICAL TRIAL: NCT04366830
Title: Intermediate-size Expanded Access of Remestemcel-L, Ex-vivo Cultured Adult Human Mesenchymal Stromal Cells for Acute Respiratory Distress Syndrome Due to COVID-19 Infection
Brief Title: Intermediate-size Expanded Access Program (EAP), Mesenchymal Stromal Cells (MSC) for Acute Respiratory Distress Syndrome (ARDS) Due to COVID-19 Infection
Status: No longer available | Type: Expanded Access
Sponsor: Mesoblast International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Other Study IDs: MSB-MSC-ARDS001
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2020-04

CONDITIONS: Moderate to Severe Acute Respiratory Distress Syndrome Associated With COVID-19
Keywords: ARDS; COVID-19; Coronavirus; MSC; remestemcel-L; Mesoblast; mesenchymal
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — remestemcel-l

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: Remestemcel-L — Participants will receive remestemcel-L in two infusions of 2 x 10^6 mesenchymal stromal cells per kilogram (MSC/kg), administered intravenously (IV).

SUMMARY:
The objectives of this intermediate-size expanded access protocol are to assess the safety and efficacy of remestemcel-L in participants with ARDS due to coronavirus infection 2019 (COVID-19).

DETAILED DESCRIPTION:
This intermediate-size expanded access protocol plans to treat approximately 50 adult participants, male and female, with moderate to severe ARDS due to COVID-19 infection. Participants who are 18 years of age or older will be enrolled at multiple clinical sites across the United States.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Participant has coronavirus disease COVID-19 confirmed by real-time reverse transcription polymerase chain reaction (RT-PCR) assay or another diagnostic test
3. Moderate to severe ARDS as determined by the following criteria (adapted from the Berlin criteria):

   * Bilateral opacities must be present on a chest radiograph or computed tomographic (CT) scan. These opacities are not fully explained by pleural effusions, lobar collapse, lung collapse, or pulmonary nodules.
   * Respiratory failure not fully explained by cardiac failure or fluid overload. An objective assessment (e.g., echocardiography) to exclude hydrostatic pulmonary edema is required if no risk factors for ARDS are present.
   * Moderate to severe impairment of oxygenation must be present, as defined by the ratio of arterial oxygen tension to fraction of inspired oxygen (PaO2/FiO2). The severity of the hypoxemia defines the severity of the ARDS:

     * Moderate ARDS: e PaO2/FiO2 >100 millimeters of mercury (mmHg) and ≤200 mmHg, on ventilator settings that include positive end-expiratory pressure (PEEP) ≥5 centimeters (cm) of water OR
     * Severe ARDS: PaO2/FiO2 ≤100 mmHg on ventilator settings that include PEEP ≥5 cm of water
4. ≤72 hours post-initiation of ventilation
5. High sensitivity C-reactive protein (hs-CRP) serum level ≥ 4.0 milligrams per deciliter (mg/dL)
6. Acute Physiologic and Chronic Health Evaluation (APACHE II) score ≥5
7. Aspartate aminotransferase/alanine transaminase (AST/ALT) < 5x upper limit of normal (ULN)
8. Creatinine clearance ≥ 30 milliliters per minute (mL/min)
9. Serum creatinine <2 mg/dL

Exclusion Criteria:

1. Participant is receiving extracorporeal membrane oxygenation (ECMO)
2. Females who are pregnant or lactating
3. Known hypersensitivity to dimethyl sulfoxide (DMSO) or to porcine or bovine proteins
4. Severe chronic obstructive pulmonary disease (COPD) requiring oxygen therapy prior to becoming ill with ARDS due to COVID-19 infection
5. Any end-stage organ disease which, in the opinion of the treating physician, may possibly affect the safety of the remestemcel-L treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Burke, ANP-C, Study Director — Mesoblast, Inc.
Locations (1):
- Mount Sinai Hospital, New York, New York, United States